CLINICAL TRIAL: NCT03079440
Title: Phase 2 Study of Temozolomide Plus Capecitabine in Patients With Grade 3 and Low Ki-67 Gastroenteropancreatic Neuroendocrine Tumors
Brief Title: TEMCAP in Grade 3 and Low Ki-67 Gastroenteropancreatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Baek-Yeol Ryoo, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Asan-ONCHBP-2017-002
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Carcinoma; Temozolomide; Capecitabine
Keywords: Neuroendocrine tumors; Neuroendocrine Carcinoma; Capecitabine; Temozolomide
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — Temozolomide; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TEMCAP (Experimental): Temozolomide plus Capecitabine
  Interventions: Drug: TEMCAP

INTERVENTIONS:
Drug: TEMCAP — Oral capecitabine 750 mg/m2 twice a day, Day 1 to 14 and oral temozolomide 200 mg/m2 once a day, Day 10 to 14
  Other Names: Temozolomide and capecitabine

SUMMARY:
GI tract including pancreas is the one of most common primary sites of neuroendocrine tumors. Current grading of neuroendocrine tumors are based on the 2010 WHO classification. This classifies grade 3 tumors as the neuroendocrine tumor with mitosis > 20 per 10 high power field or Ki-67 labeling index > 20%. Etoposide-based chemotherapy, mostly as the combination with cisplatin, has been the mainstay of the treatment for patients with grade 3 neuroendocrine tumors. However, a recent large retrospective analysis has suggested this regimen may not be effective in relatively low Ki-67 labeling index. Therefore, the investigators designed a clinical trial testing temozolomide-capecitabine combination, which has been mostly investigated in well differentiated (ie., grade 1 or 2) neuroendocrine tumors, in patients with grade 3 and low Ki-67 gastroenteropancreatic neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years and older
* Histologically confirmed neuroendocrine tumors of gastrointestinal tract or pancreas
* Unresectable or metastatic disease
* Grade 3 according to the 2010 WHO classification (Ki-67 labeling index > 20% or > 20 mitoses per 10 high power field)
* Ki-67 labeling index < 60%
* At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 ~ 2
* Adequate bone marrow function as defined by platelets ≥ 100 x 109/L and neutrophils ≥ 1.5 x 109/L
* Adequate renal function, with serum creatinine < 1.5 x upper limit of normal (ULN)
* Adequate hepatic function with serum total bilirubin < 2 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 x ULN
* No other malignant disease apart from non-melanotic skin cancer or carcinoma in situ of the uterine cervix or any other non life-threatening cancer (i.e., prostate or thyroid cancer) except where treated with curative intent > 5 years previously without evidence of relapse
* Written informed consent to the study

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol or a history of non-compliance
* Last dose of radiotherapy received within 4 weeks before the start of study treatment, excluding palliative radiotherapy
* Obstruction of gastrointestinal tract
* Active gastrointestinal bleeding
* Myocardial infarction within 6 months prior to the study medication, and other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol
* Female subjects who are pregnant or lactating, or males and females of reproductive potential not willing or not able to employ a highly effective method of birth control/contraception to prevent pregnancy from 2 weeks before receiving study drug until 3 months after receiving the last dose of study drug. A highly effective method of contraception is defined as having a low failure rate (< 1% per year) when used consistently and correctly.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Response rate | 2 years
  Proportion of patients with complete or partial response graded by Response Evaluation Criteria in Solid Tumors version 1.1

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Time between the start of study treatment and disease progression
Overall survival | 2 years
  Time between the start of study treatment and survival
Toxicity (Adverse events graded by National Cancer Institute-Common Terminology Criteria version 4.03) | 2 years
  Adverse events graded by National Cancer Institute-Common Terminology Criteria version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Baek-Yeol Ryoo, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Carbonero R, Sorbye H, Baudin E, Raymond E, Wiedenmann B, Niederle B, Sedlackova E, Toumpanakis C, Anlauf M, Cwikla JB, Caplin M, O'Toole D, Perren A; Vienna Consensus Conference participants. ENETS Consensus Guidelines for High-Grade Gastroenteropancreatic Neuroendocrine Tumors and Neuroendocrine Carcinomas. Neuroendocrinology. 2016;103(2):186-94. doi: 10.1159/000443172. Epub 2016 Jan 5. No abstract available. PMID 26731334
- [Background] Sorbye H, Strosberg J, Baudin E, Klimstra DS, Yao JC. Gastroenteropancreatic high-grade neuroendocrine carcinoma. Cancer. 2014 Sep 15;120(18):2814-23. doi: 10.1002/cncr.28721. Epub 2014 Apr 25. PMID 24771552
- [Background] Sorbye H, Welin S, Langer SW, Vestermark LW, Holt N, Osterlund P, Dueland S, Hofsli E, Guren MG, Ohrling K, Birkemeyer E, Thiis-Evensen E, Biagini M, Gronbaek H, Soveri LM, Olsen IH, Federspiel B, Assmus J, Janson ET, Knigge U. Predictive and prognostic factors for treatment and survival in 305 patients with advanced gastrointestinal neuroendocrine carcinoma (WHO G3): the NORDIC NEC study. Ann Oncol. 2013 Jan;24(1):152-60. doi: 10.1093/annonc/mds276. Epub 2012 Sep 11. PMID 22967994
- [Background] Strosberg JR, Fine RL, Choi J, Nasir A, Coppola D, Chen DT, Helm J, Kvols L. First-line chemotherapy with capecitabine and temozolomide in patients with metastatic pancreatic endocrine carcinomas. Cancer. 2011 Jan 15;117(2):268-75. doi: 10.1002/cncr.25425. Epub 2010 Sep 7. PMID 20824724
- [Background] Welin S, Sorbye H, Sebjornsen S, Knappskog S, Busch C, Oberg K. Clinical effect of temozolomide-based chemotherapy in poorly differentiated endocrine carcinoma after progression on first-line chemotherapy. Cancer. 2011 Oct 15;117(20):4617-22. doi: 10.1002/cncr.26124. Epub 2011 Mar 31. PMID 21456005